CLINICAL TRIAL: NCT06984926
Title: Safety, Tolerability and Pharmacokinetics of Multiple Rising Doses of BI 3810477 in Healthy Male and Female Trial Participants (Single-blind, Randomised, Placebo-controlled, Parallel Group Design)
Brief Title: A Study to Test How Well Multiple Doses of BI 3810477 Are Tolerated by Healthy Adults
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1530-0002; 2024-519327-20-00 (Registry Identifier: CTIS); U1111-1314-5841 (Registry Identifier: WHO International Clinical Trials Registry Platform (ICTRP))
Record Dates: First submitted 2025-05-15; First posted 2025-05-22 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- BI 3810477_dose group 1 (Experimental)
  Interventions: Drug: BI 3810477
- BI 3810477_dose group 2 (Experimental)
  Interventions: Drug: BI 3810477
- BI 3810477_dose group 3 (Experimental)
  Interventions: Drug: BI 3810477
- BI 3810477_dose group 4 (Experimental)
  Interventions: Drug: BI 3810477
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 3810477 — BI 3810477
  Arms: BI 3810477_dose group 1; BI 3810477_dose group 2; BI 3810477_dose group 3; BI 3810477_dose group 4
Drug: Placebo — Placebo for BI 3810477
  Arms: Placebo

SUMMARY:
The main objectives of this trial are to investigate safety, tolerability, and pharmacokinetics of BI 3810477 in healthy male and female trial participants when given as multiple rising doses.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female participants according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR), respiratory rate (RR), temperature), 12-lead electrocardiogram (ECG), and clinical laboratory tests.
* Age of 18 to 60 years (inclusive, to be checked at time of signing informed consent).
* BMI of 18.5 to 29.9 kg/m2 (inclusive).
* Signed and dated written informed consent in accordance with international conference on harmonization-good clinical practice (ICH-GCP) and local legislation prior to admission to the trial.
* Further inclusion criteria apply.

Exclusion Criteria:

* Any finding in the medical examination (including BP, PR, RR, temperature or ECG) deviating from normal and assessed as clinically relevant by the investigator.
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 millimetre of mercury (mmHg), diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 45 to 100 beats per minute (bpm).
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance.
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator.
* Further exclusion criteria apply.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2025-06-06 (Actual); Primary Completion 2026-03-09 (Estimated); Study Completion 2026-03-09 (Estimated)

PRIMARY OUTCOMES:
Occurrence of any treatment-emergent adverse events assessed as drug-related by the investigator | Up to Day 117

SECONDARY OUTCOMES:
Area under the concentration-time curve of BI 3810477 in plasma at steady state over a uniform dosing interval τ (AUCτ,ss) | Up to Day 117
Maximum measured concentration of BI 3810477 in plasma at steady state (Cmax,ss) | Up to Day 117

CONTACTS AND LOCATIONS:
Locations (1):
- SGS Life Science Services - Clinical Research, Edegem, Belgium

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com